CLINICAL TRIAL: NCT04366544
Title: Effects of an 8-day Advanced Meditation Samyama, on Physical, Psychological and Spiritual Well-being ,and Associated Neural Mechanisms
Brief Title: Effects of an 8-day Advanced Meditation, Samyama on Physical, Psychological and Spiritual Wellbeing ,and Associated Neural Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Senthilkumar Sadhasivam, MD, MPH, MBA, Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1801728792
Record Dates: First submitted 2020-04-17; First posted 2020-04-29 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Mental Health Wellness 1; Happiness; Depression; Consciousness, Level Altered; Ecstasy; Dietary Habits; Stress; Inflammatory Bowel Diseases
MeSH Terms: conditions — Depression; Consciousness Disorders; Feeding Behavior; Inflammatory Bowel Diseases | interventions — Medicare Part B

STUDY DESIGN:
Intervention Model Description: Potential participants will be sent email invitations approximately 2 months prior to the program. Participants will have the options to take part in online surveys, blood samples, and/or stool samples. Up to 1000 participants (attendees and spouses/significant others) may take the online surveys twice before the samyama program, 2 weeks after and 3 months after. Up to *200 may volunteer to have 4 blood draws. 150 volunteers may also send in 3 stool samples - 1. prior to starting the Samyama pre-prep diet 2. within one week of the Samyama program 3. After returning home from the program.
  Up to 50 spouses/significant others living with Samyama attendees will also be offered the opportunity to complete a shortened version of the online surveys, provide blood and/or stool samples.
  *Up to 200 volunteers at Isha can participate in blood draws. Upto 25 subjects will also be enrolled in the (2)EEG and (2)fMRI Study before and after Samyama.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time Point 1: Baseline/Pre-preparatory Samyama (Other): * Survey link for participant
  * Survey link for spouse/ "control"
  * Stool collection from home
  * Blood sample at home provided by at home phlebotomy services or at Isha Center group meditation by study personnel.
  Interventions: Other: Part A1: Survey; Other: Part A2: Sample collection
- Time point 2: Post-Preparatory/Pre-Samyama (Other): * Online Surveys
    * Participant
    * Spouse
  * Stool collection from IIIS/home
  * Blood sample collection: on site at IIIS/home EEG and fMRI
  Interventions: Other: Part A1: Survey; Other: Part A2: Sample collection; Other: Part B:
- Timepoint 3: Immediate Post-Samyama (Other): * Online survey to be completed
  * Survey link for participant
  * Survey link for spouse
  * Blood sample collection: on site at IIIS o Participant only - Not spouse/significant other. EEG and fMRI
  Interventions: Other: Part A1: Survey; Other: Part A2: Sample collection; Other: Part B:
- Timepoint 4: 3 months Post Samyama (Other): * Blood draw at home by at home phlebotomist
  * Post program online survey follow up to be completed
  * Survey link for participant
  * Survey link for spouse: https
  * Stool collection from home
  Interventions: Other: Part A1: Survey; Other: Part A2: Sample collection

INTERVENTIONS:
Other: Part A1: Survey — Online
Other: Part A2: Sample collection — Blood and Stool
Other: Part B: — EEG and fMRI
  Arms: Time point 2: Post-Preparatory/Pre-Samyama; Timepoint 3: Immediate Post-Samyama

SUMMARY:
The purpose of this study is to investigate the effects of Samyama program on blood levels of selected neurotransmitters before and after the program, and associate with corresponding effects on mind/psyche before and after the program in adult participants.

Hypothesis:

1. The state of higher consciousness and ecstasy resulting from Samyama result from increased levels of Anandamide, an endocannabinoid, and Brain Derived Neurotrophic Factor (BDNF).
2. The 60-day preparatory phase that includes dietary regulation and yogic practices will reduce the gut inflammation and thereby will improve the gut microbiome.

DETAILED DESCRIPTION:
Potential participants (those signed up to attend the Samyama program at Isha) will be sent email invitations approximately 2 months prior to the program. Participants will have the options to take part in online surveys, blood samples, and/or stool samples. Up to 1000 participants (attendees and spouses/significant others) may take the online surveys twice before the samyama program, 2 weeks after and 3 months after. Up to *200 may volunteer to have 4 blood draws. (Blood draws will occur 1. At home, or at an Isha group meditation, 1-2 months prior to Samyama 2. At Isha before the start of the program 3. At Isha after the program 4. At home after returning from the Samyama program). 150 volunteers may also send in 3 stool samples - 1. prior to starting the Samyama pre-prep diet 2. within one week of the Samyama program 3. After returning home from the program.

Up to 50 spouses/significant others living with Samyama attendees will also be offered the opportunity to complete a shortened version of the online surveys, provide (2) blood and/or (3) stool samples. Blood would be collected at home prior to their spouses/significant other's Samyama attendance and in their home after the program. Requested stool samples would be asked to be collected approximately 1 month prior to the program, 1 week prior to the program and one week after the program.

Blood samples will be sent to Indiana University and may be sent to other specialty labs for additional analysis. Genetic and future biomarker samples will be stored at the PI's Indiana University lab facilities.

If survey participants do not complete surveys during suggested time periods, they may also be sent reminders (via emails) to complete surveys.

*Only up to 150 volunteers will have at home blood draws (or blood draws at an Isha group meditation). Only those who participated in the pre-Samyama at home blood draws will be asked to participate in the post-Samyama blood draws.

Up to 200 volunteers at Isha can participate in blood draws (regardless of whether they participated in at home blood draw).

Those who complete the survey will also be asked if they have a significant other or spouse who lives with them who would be willing to complete surveys, and participate in blood draws and/or provide stool samples. Participants with willing spouses will be asked to enter an email address for that spouse/significant other. Spouse/significant other will be emailed the invitation with study information.

Upto 25 subjects will also be enrolled in the (2)EEG and (2)fMRI Study March 19 and March 29, 2018 (before Samyama), and between April 9th and May 9th, 2018 (after Samyama).

ELIGIBILITY:
Inclusion Criteria:

1. Advanced meditation program participants age 18 or older (and interested spouses/significant others who live with meditation program participants.)

Exclusion Criteria:

1. Inability to read and comprehend the consent form
2. Subjects with medical conditions in which a blood draw would be contra-indicated (e.g. severe anemia).
3. Active marijuana/opioid and related drug use
4. Probiotic or prebiotic supplements within 60 days of enrollment
5. Antibiotic use within 60 days of enrollment
6. Participants living outside of the country.
7. Spouses who indicate in the online survey that they participate in meditation will be excluded from stool and blood samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
levels of Anandamide | 4 months
  Anandamide (AEA) activates endocannabinoid-1 (eCB1) receptors in the central nervous system and eCB2 receptors throughout the body and studies have suggested its role in regulating mood and behavior, sleeping and eating patterns, memory, pain, immune system, fertility and cancer inhibition [3]. Endogenous anandamide is mainly active at eCB1 receptor, which is responsible for the experience of blissfulness, ecstasy and the elevated mood and wellbeing similar to psychoactive effects reported in cannabis use. Anandamide is thought to be related to the experience of "runner's high" due to intense physical activity [4]. So far, no study has explored the effect of yoga and meditation on endogenous levels of anandamide in humans. However, Anandamide is very quickly catabolized in the human system by Fatty Acid Amide Hydrolase (FAAH) [5]. So, to control for this we propose to use FAAH inhibitor in the sampling tube to preserve and accurately measure anandamide.
Levels of Brain Derived Neurotrophic Factor (BDNF) | 4 months
  Brain-derived neurotrophic factor (BDNF) is another neurotransmitter found in the brain and the rest of the body. It helps in survival of existing neurons and growth of new neurons. It is involved in regulation of other neurotransmitters, long-term memory, stable memory function and cognitive function [6, 7]. Studies have suggested negative correlations between BDNF levels and disease such as depression, schizophrenia, obsessive-compulsive disorder, Alzheimer's disease, anorexia and dementia. Studies have shown beneficial increase in BDNF levels in human subjects because of yoga and meditation practices [8].
Transcriptome analysis | 4 months
  Transcriptome analysis (RNA sequencing - gene expression analyses): Peripheral blood from participants will be collected before and after Samyama in PAXgene Blood RNA Tubes (Qiagen). Upon RNA extraction, RNA quantity will be assessed with Nanodrop (Nanodrop Technologies) and quality with the Agilent Bioanalyzer (Agilent Technologies). RNA samples will be cleaned using DNAse I kit according to the Rapid out removal DNA kit instruction (Thermoscientific) and will be converted into cDNA by using Lexogen QuantSeq 3' Fwd Library Prep Kit (Lexogen) according to manufacturer's instruction to generate compatible library for Illumina sequencing. cDNA libraries will be assessed using TapeStation (Agilent Technologies, USA) before 65-100 bp single end sequencing using Illumina HiSeq 4000 system based on standard protocols to obtain raw sequencing data. Raw sequencing reads will be processed using our standard pipelines to obtain high quality sequencing reads for data analyses.
Epigenetic analysis (DNA methylation) | 4 months
  Epigenetic analysis (DNA methylation): DNA from peripheral blood of participants will be examined for integrity by agarose gel electrophoresis and quantified using fluorimeter using a double stranded DNA (BR) assay (Thermo Fisher Scientific). About 500 ng of the sampled DNA will be analyzed on a Infinium® MethylationEPIC BeadChip (Illumina, San Diego, CA). The hybridized and stained arrays will be ultimately scanned using HiScanSQ system (Illumina). Infinium MethylationEPIC (EPIC) BeadChip from Illumina will evaluate over 850,000 methylation sites quantitatively across the genome at single-nucleotide resolution. Data analyses will be performed utilizing previously published standard pipelines.

SECONDARY OUTCOMES:
Microbiome analysis: | 4 months
  Microbiome analysis: Participants will also be requested for stool samples prior to, or early into the start of preparatory steps (approximately 60 days before the scheduled program start), within 2.5 weeks prior to the program, and another one after the completion of the program. The strict vegan diet and the preparatory steps along with the Samyama meditation program is hypothesized to reduce the gut inflammation and improve the gut microbiome.
Gut Inflammation analysis: | 4 months
  Gut Inflammation analysis: We will explore the relations between perceived stress, blood cortisol, plasma tryptophan catabolites (i.e., kynureine and quinolinic acid), and cytokines potentially related to UC (GM-CSF, Eotaxin, IFN-α, IP-10, IFN-γ, MCP-1, IL-1β, MIG, IL-1RA, MIP-1α, IL-2, MIP-1β, IL-2R, RANTES, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12 (p40/p70), IL-13, IL-15, IL-17, and TNF-α)
Plasma lipidomic analyses: | 4 Months
  Plasma lipidomic analyses: A high-resolution (0.2 to 3 ppm mass error) mass spectrometric, non-targeted lipidomics platform will be utilized to compare the plasma lipidome of Samyama participants before and after the program. Blood samples will be collected at the following three time points: (1) before the start of the Samyama program, (2) after the Samyama program, and (3) possibly at 3 months after the program.

OTHER OUTCOMES:
fMRI | 4 months
  fMRI: Functional MRI is a useful non-invasive tool to study brain neuronal activity.
  Examine the qualitative fMRI changes associated with 8-day advanced meditation, Samyama program. This would specifically examine the resting state neuroconnectivity, in particular the 'default mode network'. Anatomical changes such as grey matter volume and insular thickness will also be analyzed. fMRI changes with meditative breath watching will also be recorded and analysed.
EEG | 4 months
  EEG: Studies have shown that EEG can be used to explore the temporal relation between measures of functional connectivity network integration and meditation quality. van Lutterveld et al studied the functional connectivity with the help of Minimum spanning tree (MST) and graph measures.
  Examine the EEG changes associated with 8-day advanced meditation, Samyama program.

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
MRI and EEG data from Indiana University and a collaboring site, part of Harvard University will be combined to increase the statistical power. De-identified MRI and EEG data will be mutually shared with Boston investigators (PI: Dr. Balachundhar Subramaniam).
Supporting Information: Study Protocol, SAP
Time Frame: Until the data is completely analyzed
Access Criteria: Deidentified

REFERENCES:
- [Derived] Raman M, Vishnubhotla R, Ramay HR, Goncalves MCB, Shin AS, Pawale D, Subramaniam B, Sadhasivam S. Isha yoga practices, vegan diet, and participation in Samyama meditation retreat: impact on the gut microbiome & metabolome - a non-randomized trial. BMC Complement Med Ther. 2023 Apr 5;23(1):107. doi: 10.1186/s12906-023-03935-8. PMID 37020274
- [Derived] Vishnubhotla RV, Wood PL, Verma A, Cebak JE, Hariri S, Mudigonda M, Alankar S, Maturi R, Orui H, Subramaniam B, Palwale D, Renschler J, Sadhasivam S. Advanced Meditation and Vegan Diet Increased Acylglycines and Reduced Lipids Associated with Improved Health: A Prospective Longitudinal Study. J Integr Complement Med. 2022 Aug;28(8):674-682. doi: 10.1089/jicm.2022.0480. Epub 2022 May 9. PMID 35532984
- [Derived] Vishnubhotla RV, Radhakrishnan R, Kveraga K, Deardorff R, Ram C, Pawale D, Wu YC, Renschler J, Subramaniam B, Sadhasivam S. Advanced Meditation Alters Resting-State Brain Network Connectivity Correlating With Improved Mindfulness. Front Psychol. 2021 Nov 18;12:745344. doi: 10.3389/fpsyg.2021.745344. eCollection 2021. PMID 34867626

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/44/NCT04366544/Prot_SAP_000.pdf